CLINICAL TRIAL: NCT07376616
Title: Cardiovascular Research in EMbarazo and MAternity (EMMA). Study on Heart Rate Variability and Hemodynamic Adaptations During Pregnancy and Postpartum.
Acronym: EMMA
Status: Recruiting | Type: Observational
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Sponsor
Other Study IDs: EMMA
Record Dates: First submitted 2025-12-12; First posted 2026-01-29 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy Related; Heart Rate Variation (HRV); Hemodynamics
MeSH Terms: interventions — Blood Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Unic group
  Interventions: Other: Assessment of HRV and blood pressure

INTERVENTIONS:
Other: Assessment of HRV and blood pressure — Assessment of Heart Rate Variation (HRV) and blood pressure

SUMMARY:
Heart rate variability (HRV) provides a non-invasive assessment of autonomic control of the nervous system over the heart. During pregnancy, the cardiovascular system adapts significantly, affecting HRV and hemodynamics. Studying the relationship between HRV and hemodynamic changes is critical to understanding and monitoring cardiovascular health during pregnancy and postpartum, and predicting potential complications.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Pregnancy from the third month of gestation
* No pre-existing cardiovascular disease
* Good cognitive level
* Sign informed consent

Exclusion Criteria:

* Diabetes mellitus
* Hyperthyroidism
* Hypothyroidism
* Chronic hypertension diagnosed before pregnancy
* Heart failure
* Ischemic heart disease or malignant ventricular arrhythmias (ventricular fibrillation, ventricular tachycardia, grade 2 or 3 AV block, atrial fibrillation in patients with Wolff-Parkinson- White syndrome, paroxysmal fibrillation or flutter with rapid ventricular response and hemodynamic deterioration, uncontrolled supraventricular tachycardia)
* Exercise-induced ischaemia
* Unstable angina
* Disease not susceptible to revascularization
* Associated valvular heart disease
* Chronic kidney disease
* Degenerative neurological condition
* Brain aneurysms
* Arteriovenous malformations
* History of transient cerebral infarction (ICTUS)
* Migraines diagnosed
* Epilepsy
* Brain or spinal cord injury
* Tumors
* Diseases of the respiratory tract
* Diseases of lung tissue
* Diseases of pulmonary circulation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women pregnant from the first trimester of gestation over 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
RR (R-R range) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  The RR interval is the time between successive R-waves of the QRS complex now electrocardiogram (ECG) expressed in milliseconds (ms). It is a fundamental unit in HRV analysis and represents the time between two consecutive heartbeats.
RMSSD (Root Mean Square of Successive Differences) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  RMSSD is a measure in the tempo domain that quantifies variability in the length of consecutive RR intervals expressed in milliseconds (ms). It reflects short-term HRV and is influenced by the parasympathetic nervous system.
pNN50 (Percentage of successive RR intervals differing by more than 50 ms) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  pNN50 is another measure in the time domain that represents a percentage (%) of RR intervals that differ by more than 50 ms. It is also indicative of short-term HRV and is related to parasympathetic activity.
HF (High Frecuency) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  HF is a measurement in the frequency domain that represents the power of heart rate variability in the high frequency range (typically 0.15 to 0.4 Hz). It is associated with parasympathetic (vagal) activity and is often analyzed by spectral analysis of the HRV signal. Expressed in milliseconds squared (ms^2).
LF (low frequency) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  LF is a measurement in the frequency domain that represents the power of heart rate variability at low frequencies (usually from 0.04 to 0.15 Hz). The LF is influenced by sympathetic and parasympathetic activity and the child analyzase xunto coa IC. Expressed in milliseconds to frame (ms^2).
SD1 (standard deviation 1) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  SD1 is xeometric measures derived from Poincaré graphs, which are graphical representations of RR intervals. SD1 represents the short-term variability perpendicular to the identity line in the Poincaré graphic and is influenced by parasympathetic activity.
SD2 (standard deviation 2) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  SD2 is a xeometric measure derived from Poincaré graphs, which are graphical representations of RR intervals. SD2 represents long-term variability along the identity line and is influenced by sympathetic and parasympathetic activity.
DFAa1 (Trend Flotation Analysis, alpha-1) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  DFA is a mathematical method used to evaluate fractal properties in time series, such as the HRV. DFAa1 centrase specifically in short-term floatation (alpha-1) in the HRV signal. It offers information about the properties of autosemellanza or long-range correlation of the signal.
DFAa2 (Trend Flotation Analysis, alpha-2) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  DFA is a mathematical method used to evaluate the fractal properties of time series, such as HRV. DFAa2 céntrase especially in long-term flotation (alpha-2) in the HRV signal.
SampEn (Sample Entropy) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  The show entropy is a modified algorithm less dependent on the duration of the time series. Used to evaluate the complexity of R-R intervals. A higher entropy value represents more complex dynamics and greater ability of the cardiovascular system to adapt to changes, which is associated with lower cardiovascular health.
ApEn (approximate entropy) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  ApEn is a measure used to evaluate the regularity and complexity of time series, such as HRV. ApEn quantifies the degree of unpredictability in the time series fluctuations, providing information about the structure of the signal and its irregularity. A lower value of ApEn indicates a more regular and predictable series, whereas a higher value reflects greater complexity and irregularity.
MSE (Multiscale entropy) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  MSE is an extension of SampEn that analyzes the complexity of time series on multiple time scales. The MSE allows to evaluate the structure of the signal at different levels of detail, providing a more complete view of its complexity.
D2 (Correlation dimension) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  The correlation dimension is a measure that estimates the minimum number of variables needed to build a model of the dynamics of a system. The greater the number of variables required to predict a time series, the greater its complexity. This measure provides information about the subcomplex and dynamic characteristics of the system.
Heart rate turbulence (HRT) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  The cardiac frequency turbulence and a baroreflex-mediated axus of the cardiac frequency that acts as a countermechanism for premature ventricular contraction. It consists of no brief acceleration of the heart rate, followed by a slow decrease at the reference rate.
Heart rate (HR) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  Number of heartbeats per minute during treatments performed during different trimesters of pregnancy and not postpartum (Lat/min).
Systolic blood pressure (PAS) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  Perform a systolic blood pressure record expressed in mmHg and measured in different locations.
Diastolic blood pressure (DBP) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  Perform a diastolic blood pressure record expressed in mmHg and measured in different locations.
Mean arterial pressure (MAP) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  MAP is the constant blood pressure value that, wedge same peripheral resistance would produce the same flow rate (minute cardiac volume) as xera a variable blood pressure (systolic and diastolic pressure) expressed in mmHg.
Pulse pressure (BP) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  BP is an index of arterial distensibility expressed in mmHg obtained from the difference between systolic and diastolic blood pressure and measured in different locations.
O2 saturation | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  Oxygen saturation measures, in different locations, the percentage of hemoglobin in red blood cells currently transporting oxygen, indicating how well the lungs and heart are oxygenating body tissues.
Cardiac output (CO) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  Cardiac output is the total volume of blood pumped by the heart's left ventricle in one minute, serving as a critical indicator of cardiovascular health and tissue perfusion. It is measured in L/min
Stroke volume (SV) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  Stroke volume is the volume of blood pumped from the left ventricle per beat. It is measured in mL
Vascular resistance | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  Vascular resistance is the opposition to blood flow caused by friction between blood and vessel walls. It is measured in dyn*s/cm^5
Cerebral vascular flow | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  Cerebral blood flow (CBF) is the net amount of blood delivered to the brain's capillary bed per unit of time and tissue mass, typically measured in mL/min/100g
Cardiac Index (CI | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  The Cardiac Index is a hemodynamic parameter representing the heart's pumping efficiency, calculated as the cardiac output divided by the body surface area. It measures blood flow (liters per minute) relative to a person's size L/min/m^2
PEP (Pre-Ejection Period) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  The PEP (Pre-Ejection Period) in hemodynamics is a parameter measured in milliseconds (ms) that evaluates the time that elapses from the beginning of the electrical activation of the ventricle until the beginning of the ejection of blood towards the aorta.
Ejection Time (ET) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  Ejection Time (ET) is the duration of systolic flow, measuring (in milliseconds) the time interval from aortic valve opening to closure when the left ventricle ejects blood into the aorta.
Maternal ultrasound | Pregnancy weeks 13, 27 and 41.
  Maternal ultrasound allows obtaining multiple biometric (measurements) and morphological (structures) variables that are fundamental to evaluating fetal development, maternal well-being, and gestational age.

SECONDARY OUTCOMES:
Age | Basal assessment
  Age expressed in years
Race | Basal assessment
  Caucasian, Black or of African descent, Arab or North African, Asian, Native American, Latin American, Other
Births | Basal assessment
  Nulliparous, primiparous, multiparous
Fertilization | Basal assessment
  Spontaneous, Conventional IVF, ICSI, FET (frozen embryos), Mini IVF, Ovodonation, ROPA Method
Risk of pre-eclampsia | Basal assessment
  High, Medium, Low
Previous pregnancies | Basal assessment
  Number of pregnancies
Previous spontaneous abortions | Basal assessment
  Number of pregnancies
Type of childbirth | Basal assessment
  Spontaneuos vaginal, assisted vaginal, scheduled cesarean, urgent cesarean
Time of childbirth | Basal assessment
  Pre-term, at term, post-term
Level of education | Basal assessment
  No studies, primary education, secondary, baccalaureate, vocational training, university studies
Employment status | Basal assessment
  Full-time paid employment, part-time paid employment, self employed, unemployed, dedication to the home
Concomitant medication | Basal assessment
  Without medication, Analgesics, Antibiotics, Antivirals, Antifungals, Antiparasitics, Anti-inflammatory drugs, Antihistamines, Antihypertensive drugs, Hypoglycemic agents, Antidepressants, Anxiolytics, Antipsychotics, Diuretics, Anticoagulants, Nutritional supplementation, Antiemetics, Hormone treatment before pregnancy, Hormone treatment in pregnancy, Other
Smoking habit | Basal assessment
  Non-smoker, Ex-smoker more than one year, Ex-smoker less than a year, Non-smoker during pregnancy, Smoker
Consumption of alcohol | Basal assessment
  Non-consumer, Ex-consumer, Not consuming during pregnancy, Occasional consumer, Daily consumer
Family history of disease | Basal assessment
  No background, High blood pressure, Type 2 diabetes mellitus (T2DM), Hypertensive disorders during pregnancy, Other
Weight | Basal assessment
  Kg
Height | Basal assessment
  Cm
Pregnancy-associated plasma A protein (PAPP-A) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  Biomarker of preeclampsia expressed in MoM
Placental growth factor (PlGF) | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  Biomarker of preeclampsia expressed in pg/mL
Ratio sFlt-1/PlGF | Pregnancy weeks 13, 27 and 41. Postpartum month, 3, 6 and 12 months.
  Biomarker of preeclampsia
Postpartum physical activity habits (IPAQ) | Postpartum month, 3, 6 and 12 months.
  Low, moderate, high
Physical activity habits in pregnancy (PPAQ) | Pregnancy weeks 13, 27 and 41
  METS-h/week
Postpartum specific anxiety scale (PSAS - ES) | Postpartum month, 3, 6 and 12 months.
  Minimal anxiety, Mild anxiety, Moderate anxiety, Severe anxiety
Edinburgh Scale for Postnatal Depression (EPDS - ES) | Postpartum month, 3, 6 and 12 months.
  No postnatal depression, Mild symptoms, Moderate symptoms, Significant symptoms
Maternal-fetal complications in pregnancy | Pregnancy weeks 13, 27 and 41
  No complications, Severe nausea and vomiting, Pre-eclampsia, Gestational hypertension, Gestational diabetes, Infections, Anemia, Detachment of placenta, Restriction of intrauterine growth, Placenta previa, Other
Postpartum complications | Postpartum month, 3, 6 and 12 months.
  No complications, Postpartum hypertension, Postpartum hemorrhage, Postpartum infections, Postpartum depression, Deep vein thrombosis or pulmonary embolism, Perineal pain, Other
Hospitalizations pregnancy | Pregnancy weeks 13, 27 and 41
  Number
Reason hospitalization | Pregnancy weeks 13, 27 and 41
  No hospitalization, Severe nausea and vomiting, Infections, Abnormal vaginal bleeding, Postpartum bleeding, Postpartum infections, Complications from cesarean section, Mood disorders, Cardiorespiratory complications, Other

CONTACTS AND LOCATIONS:
Overall Officials: Alicia González Represas, Principal Investigator — Instituto de Investigación Sanitaria Galicia Sur (IISGS)
Locations (1):
- Hospital Alvaro Cunqueiro, Vigo, Pontevedra, Spain